CLINICAL TRIAL: NCT00596206
Title: Assessment of the Early Efficacy Response Rate of Leflunomide According to the Initial Dosing Regimen in the Treatment of Naive-DMARD (Disease Modifying Anti-Rheumatic Drug) Early RA (Rheumatoid Arthritis)-Patients
Brief Title: Leflunomide EfficAcy Response Related to Dosing Regimen in Early Rheumatoid Arthritis
Acronym: LEADER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEFLU_R_01143; Eudract#: 2007-000886-40
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 100 mg of leflunomide
  Interventions: Drug: leflunomide
- 2 (Active Comparator): 20 mg of leflunomide
  Interventions: Drug: leflunomide

INTERVENTIONS:
Drug: leflunomide — 20 or 100 mg per os, Film coated tablet, for 3 days + matching placebo, then 20 mg once daily for 3 months

SUMMARY:
To assess the efficacy response rate at 3-months of two dosing regimen of leflunomide in DMARDs-naive patients presenting an early-RA using American College of Rheumatology 20% response rate.

To assess the clinical efficacy at 1-month and 3-month using complementary efficacy criteria (ACR 50, ACR 70, DAS 28) in each group of treatment, To assess the clinical and biological safety using standard blood monitoring, TEAED and SAE in each group of treatment, To evaluate treatment modifications; particularity leflunomide and concomitant use of AINS and corticoids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active rheumatoid arthritis in the previous 6 months (according to the ACR guidelines)
* Must have active disease to be initiated by DMARDs (Disease Modifying Anti-Rheumatic Drugs)

Exclusion Criteria:

* Patient presenting or having a history of other inflammatory joint disease
* Patient with ongoing or previous Stevens-Johnson syndrome, toxic epidermal necrolysis or erythema multiforme
* Patient with significantly impaired bone marrow function or significant anaemia, leucopenia or thrombocytopenia due to causes or other than active rheumatoid arthritis
* Persistent infection or severe infection within 3 months before enrollment,
* Uncontrolled hypertension, uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, terminal illness or other medical condition which, in the opinion of the investigator, would put the patient at risk to participate in the study,
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Severe hypoproteinemia (e.g., in case of severe liver disease or nephrotic syndrome) with serum albumin < 3.0 g/dl
* Moderate or severe impairment of renal function, as known by serum creatinine > 133 mcmol/L (or 1.5 mg/dl)
* Patient with history of recent and clinically significant drug or alcohol abuse
* Impairment of liver function or persisting ALT (SGPT) elevations of more than 2-fold the upper limit of normal
* Pregnancy
* Breastfeeding
* Women of childbearing potential, except if they fulfill specific conditions,
* Men wishing to father children during the course of the study or within the 24 months thereafter (or 3 month with the washout procedure)
* Patient with a congenital or acquired severe immuno-deficiency, a history of cancer or lymphoproliferative disease, or any patient who has received total lymphoid irradiation
* Known HIV positive status
* Known positive serology for hepatitis B or C
* Patient with hypersensitivity to any of the excipients in the tablets of leflunomide
* Previous therapy at any time with:

  * any DMARD including methotrexate, oral or injectable gold salts, chloroquine, hydroxychloroquine, ciclosporin, azathioprine, methotrexate, sulfasalazine
  * D penicillamine
  * alkylating agents, e.g., cyclophosphamide, chlorambucil, biological agents, e.g., interferon, monoclonal antibodies, growth factor, cytokines
  * any investigational drug
  * any antimetabolites
  * any opiates
* Therapy within the previous 4 weeks with:

  * oral corticosteroids exceeding a prednisolone equivalent of 10 mg/day
  * parenteral or intra-articular corticoid injection

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy response rate using ACR 20 criteria in each initial dosing regimen group | at 3 month

SECONDARY OUTCOMES:
Clinical efficacy response rate using ACR 50, ACR 70, DAS 28 efficacy criteria in each group of treatment | at 1 and 3 months
Clinical and biological safety using standard blood monitoring, TEAED and SAE in each group of treatment | From the Informed Consent Form (ICF) signature to the end of the study
Measure of acute phase response (ESR, CRP) | At 1 and 3 months
Patient and physician global assessment | At 1 and 3 months
SF-36 questionnaire | At 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Seoul, South Korea

REFERENCES:
- [Derived] Cutolo M, Bolosiu H, Perdriset G; LEADER Study Group. Efficacy and safety of leflunomide in DMARD-naive patients with early rheumatoid arthritis: comparison of a loading and a fixed-dose regimen. Rheumatology (Oxford). 2013 Jun;52(6):1132-40. doi: 10.1093/rheumatology/kes321. Epub 2013 Feb 11. PMID 23401601